CLINICAL TRIAL: NCT02132455
Title: The Utility of Timed Segmental Withdrawal During Screening Colonoscopy for Increasing Adenoma Detection Rate. A Randomized Controlled Clinical Trial
Brief Title: The Utility of Timed Segmental Withdrawal During Screening Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Marc Zuckerman, Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: E14017
Record Dates: First submitted 2014-01-02; First posted 2014-05-07 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Colonoscopy
Keywords: Screening colonoscopy; Surveillance colonoscopy
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- 3 minutes in the right side colon (Experimental): Colonoscopy, at least 3 minutes in the right side colon from the total withdrawal time
  Interventions: Procedure: colonoscopy
- 4 minutes in the right side colon (Experimental): Colonoscopy, at least 4 minutes in the right side colon from the total withdrawal time
  Interventions: Procedure: colonoscopy
- 6 minutes whole withdrawal time (No Intervention): Colonoscopy, at least 6 minutes whole withdrawal time regardless of time spent in any segment
- 8 minutes whole withdrawal time (Experimental): Colonoscopy, at least 8 minutes whole withdrawal time regardless of time spent in any segment
  Interventions: Procedure: colonoscopy

INTERVENTIONS:
Procedure: colonoscopy — colonoscopy (colon examination with flexible tube and a camera) is to find early precancerous growth in the colon (polyps) and remove them before they turn into cancer
  Arms: 3 minutes in the right side colon; 4 minutes in the right side colon; 8 minutes whole withdrawal time

SUMMARY:
The purpose of colonoscopy (colon examination with flexible tube and a camera) is to find early precancerous growth in the colon (polyps) and remove them before they turn into cancer. The doctor performing the procedure will first advance the colonoscope to the end of the colon (cecum) and then he will examine the colon for polyps while he is withdrawing the colonoscope. The period of time that the doctor spent examining the colon called "withdrawal time". Usually doctors will spend at least 6 minutes examining the colon after he reached the cecum. The investigators are proposing that dedicating half of the withdrawal time during colonoscopy in examining the right side of the colon, will increase the detection of polyps in the right side of the colon.

DETAILED DESCRIPTION:
Research design: This is a prospective, randomized trial comparing the ADR between patients undergoing a screening colonoscopy in four different groups: 1) at least 3 minutes from the total withdrawal time dedicated to the right side of the colon, 2) at least 4 minutes from the total withdrawal time dedicated to the right side of the colon, 3) 6 minutes total withdrawal time regardless of time spent in any segment, 4) 8 minutes total withdrawal time regardless of the time spent in any segment. Randomization will be done in blocks after stratification. Four gastroenterologists and two fellows matched base on similar ADR and stratified on each arm of the study (segmental versus non-segmental withdrawal) will be performing the procedures. The estimated sample size of the four arms of the study is 400 patients.

ELIGIBILITY:
Inclusion Criteria:

* adults undergoing colonoscopy for screening or surveillance purposes

Exclusion Criteria:

* prior history of colonic surgeries
* Crohn's colitis or ulcerative colitis
* prior history of colon cancer
* poor bowel preparation
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Polyp detection rate (PDR) and Adenoma detection rate (ADR) of patients undergoing a screening colonoscopy either with segmental withdrawal protocol or with non-segmental withdrawal protocol. | 30 minutes
  Compare polyp detection rate (PDR) and ADR between patients undergoing a screening colonoscopy with segmental withdrawal protocol and with non-segmental withdrawal protocol.
The Polyp detection rate( PDR) and Adenoma detection rate (ADR) of patients undergoing screening colonoscopy either with 6-minutes or 8-minutes protocols of the segmental withdrawal. | 30 minutes
  Compare PDR and ADR between patients undergoing a screening colonoscopy with at least 6-minutes protocol versus at least 8-minutes protocol within each segmental and non-segmental withdrawal protocol.

SECONDARY OUTCOMES:
The polyp detection rate( PDR) and Adenoma detection rate (ADR) of patients undergoing screening colonoscopy either with 3-minutes or 4-minutes protocols of the non segmental withdrawal | 30 minutes
  1. Compare PDR and ADR associated with different withdrawal times with segmental and non segmental withdrawal protocol. Compare sessile serrated lesion detection rate between patients undergoing a screening colonoscopy with segmental and non segmental withdrawal protocol.
Complication rate | 1 month
  The complication rate of patients undergoing a screening colonoscopy with segmental and non segmental withdrawal protocol will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Marc Zuckerman, MD, Principal Investigator — Texas Tech University Health Science Center El Paso
Locations (1):
- Texas Tech University Health Science Center El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No